CLINICAL TRIAL: NCT05763108
Title: Clinical Significance and Coexistence of Polymorphisms of Individual Collagen-coding Genes - rs1800012 of the COL1A1 Gene and rs12722 of the COL5A1 Gene in Patellar Instability in Children.
Brief Title: Clinical Significance and Coexistence of Polymorphisms of Individual Collagen-coding Genes
Status: Completed | Type: Observational
Sponsor: Polish Mother Memorial Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PMMHRI-2021.2/1/7-GW
Record Dates: First submitted 2023-02-28; First posted 2023-03-10 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2022-10

CONDITIONS: Ligament; Laxity; Recurrent Patellar Dislocation
MeSH Terms: conditions — Joint Instability; Patellar Dislocation | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample or oral epithelial swab.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Recurrent patellar dislocation group: 50 patients with recurrent patellar dislocation and without any genetic disorders.
  Interventions: Diagnostic Test: genetic test; Other: Beighton joint laxity test
- Patients without joint hipermobility: 200 patients without recurrent patellar dislocation and genetic disorders.
  Interventions: Diagnostic Test: genetic test; Other: Beighton joint laxity test

INTERVENTIONS:
Diagnostic Test: genetic test — COL1A1 or COL5A1 genetic test
Other: Beighton joint laxity test — Based on Beighton scale.

SUMMARY:
The purpose of this study is to assess correlation between recurrent patella dislocation and genetic polymorphism rs1800012 of the COL1A1 Gene and rs12722 of the COL5A1 Gene.

DETAILED DESCRIPTION:
After being informed about the study and potential risk all of participants were performed phisical examination and genetic test. In the study we established two groups: In first group- 50 patients with recurrent patellar dislocation and without any genetic disorders. In the second one 200 patients without recurrent patellar dislocation and genetic disorders. All pediatric patients were between 7 and 17 years old in two groups respectivly.

ELIGIBILITY:
Inclusion Criteria:

• First-time diagnosed or recurrent patellar dislocation patient from 7 to 17 age years old.

Exclusion Criteria:

* Patient's age under 7.
* Presence of genetic diseases such as: Down's syndrome or Marfan's syndrome.
* Metabolic disorders.
* Previous knee surgeries.
* Cartilage and bone fractures in the knee.
* No consent for examination from the legal guardian.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients between 7 and 17 years old with recurrent dislocation of the patella without genetic diseases.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Patients with recurrent patellar dislocation | 2022-2023
  Patients with recurrent patellar dislocation
Control group without obvious joint hipermobility | 2022-2023
  Control group without obvious joint hipermobility

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof Małecki, Principal Investigator — PMMHRI
Locations (1):
- Krzysztof Małecki, Lodz, Lodzkie Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided